CLINICAL TRIAL: NCT00806325
Title: Clinical Factors Associated With the Development of Severe Sepsis in Patients Being Treated for Acute Myeloid Leukemia
Acronym: AML
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Naeem Ali, MD, Associate Professor of Medicine, Ohio State University
Other Study IDs: 2006C0052
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Sepsis; Acute Myeloid Leukemia
Keywords: Severe Sepsis; Acute Myeloid Leukemia; Sepsis in patients being treated for Acute Myeloid Leukemia
MeSH Terms: conditions — Sepsis; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — baseline blood sample drawn (2 tablespoons or 30 ml) at the beginning of the study. If subjects experience a fever another blood sample (10 ml up to 2 times) will be drawn at that time.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AML: Adult patients with AML admitted for treatment of the same

SUMMARY:
Acute leukemia is a life threatening illness that strikes people of all ages. In addition to surviving the direct effects of the disease, the treatment of leukemia generally requires chemotherapy which has its own burden. Infection is one of the most common secondary problems faced by these patients. Simple infections are common and easily treated with aggressive antibiotics. However, treated progressive infection leads to loss of vital organ function and is termed severe sepsis. Severe sepsis is associated with increased risk of death and the need for specialized care in the intensive care unit.

Besides the appropriate use of antibiotics, little is known about what clinical and patient factors are associated with the development of severe sepsis. Recent evidence has suggested that certain practices like frequent transfusion of blood products and control of glucose levels effects outcome in critically ill patients. In addition, there have been advances in our knowledge of certain genes that may predispose people to severe infections. It is possible that these factors are important in people who are not yet critically ill, but are at risk for the development of severe sepsis.

This observational study will look at genetic, clinical and therapeutic factors that are associated with the development of severe sepsis. This will help doctors understand what treatments may be helpful in preventing this serious complication.

DETAILED DESCRIPTION:
Primary hypothesis: Hyperglycemia during inpatient therapy of AML is associated with increased mortality (fewer hospital free days to Day 60, see below).

* H1a: Hyperglycemia will result in an increased risk of developing clinical signs of infection (fever).
* H1b: Hyperglycemia will be associated with an increased risk of developing severe sepsis after the onset of clinical signs of infection (fever).

  o H1b1: Hyperglycemia will be associated with the development of acute lung injury after the onset of signs of infection (fever).
* H1c: Hyperglycemia will be associated with an increased risk of ICU admission.

  o H1c1: Hyperglycemia will be associated with an increased risk of ICU admission for severe sepsis.
* H1d: Hyperglycemia will be associated with an increased risk of death in those subjects with severe sepsis (fewer hospital free days to Day 60, see below).

Secondary Aim: To investigate whether TSP-1 is important in modulating the course of sepsis-induced acute lung injury.

Secondary hypothesis: In patients with sepsis, increased levels of functional TSP-1 will be associated with a lower incidence of and a less severe course of lung injury.

* H2a: In human sepsis, increased TSP-1 levels will be associated with a lower incidence of lung-injury.
* H2b: In human sepsis, increased TSP-1 levels will be associated with a less severe course of lung-injury.
* H2c: In human sepsis, patients with the Asn682Ser polymorphism in the TSP-1 gene will be associated with a higher incidence of lung-injury.
* H2d In human sepsis, patients with the Asn682Ser polymorphism in the TSP-1 gene will be associated with a more severe course of lung-injury.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of acute myeloid leukemia
* Age ≥ 18 years of age
* Plans to receive chemotherapy as an inpatient and remain inpatient until hematologic recovery as determined by the primary treating physician

Exclusion criteria:

* Subject is unlikely to survive > 3 months with treatment
* Current diagnosis of severe sepsis
* Subject or surrogate is unable to give informed consent
* Subject is incarcerated
* Patient's family, physician, or both not in favor of endotracheal intubation or mechanical ventilation for any length of time or the presence of an advanced directive to withhold the same.
* Subject currently requiring mechanical ventilation
* Subject with current diagnosis of acute lung injury or ARDS (bilateral infiltrates on chest X-ray and PF ratio< 300 with no evidence of left atrial hypertension)
* Subject has received chemotherapy for the treatment of AML > 96 hours ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: university hospital intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
determine the true relationship of hyperglycemia to the development of severe sepsis after chemotherapy for AML | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Naeem A Ali, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No